CLINICAL TRIAL: NCT06797232
Title: "The Effect of Body Awareness Level on Shoulder Functionality and Psychological Factors in Rotator Cuff Pathologies"
Brief Title: The Effect of Body Awareness Level on Shoulder Functionality and Psychological Factors in Rotator Cuff Pathologies
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ozlem Gorgulu Goksu, PT, Msc, Medipol University
Other Study IDs: ozlemgorgulugoksu
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Syndrome
Keywords: Body Awareness Body İmage Rotator cuff Mental health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rotator Cuff Group: "A total of 25 participants aged 30-65 years with rotator cuff tendinopathy who meet the inclusion criteria, along with 25 healthy volunteers of the same age and gender, will be included."
- Healthy Group: "A total of 25 participants aged 30-65 years with rotator cuff tendinopathy who meet the inclusion criteria, along with 25 healthy volunteers of the same age and gender, will be included."

SUMMARY:
Rotator cuff syndrome is a prevalent musculoskeletal condition and the most common cause of shoulder pain. It typically begins with tendonitis and may progress to partial or complete tendon rupture due to subacromial space narrowing or overuse. Its incidence increases with age and is more common in women, often resulting in significant functional loss, reduced shoulder mobility, and lower quality of life. Shoulder pain leads to limitations in daily activities and can trigger kinesiophobia, or fear of movement, further exacerbating physical and psychological impairments.

In addition to physical limitations, individuals with rotator cuff syndrome often experience psychological challenges such as stress, anxiety, and depression. Psychological resilience-a factor influencing general well-being-plays a critical role in coping with chronic pain. High psychological resilience is associated with reduced pain severity, better shoulder functionality, and lower levels of kinesiophobia. Kinesiophobia, in turn, can lead to movement avoidance, muscle disuse, and further deterioration in function.

Basic body awareness (BBA), defined through both experiential and movement dimensions, involves understanding how the body functions and interacts with the environment. It is shaped by multiple sensory systems including proprioception, interoception, and exteroception. Body awareness is linked to pain perception, functional movement, and health-related quality of life.

Although BBA has been studied in stroke, mental health, and chronic pain, its role in shoulder rehabilitation has not been sufficiently explored. This study aims to investigate the relationship between basic body awareness, shoulder functionality, and psychological factors in individuals with rotator cuff syndrome.

DETAILED DESCRIPTION:
Rotator cuff syndrome is one of the musculoskeletal system disorders that covers a wide area. It is the most common cause of shoulder pain. The acute process begins with tendonitis of the tendons and can lead to partial rupture, degenerative changes, and eventually complete rupture. Its etiology is multifactorial, with the narrowing of the subacromial space or excessive use of the tendon being the main mechanisms. The lifetime incidence of shoulder pain observed in the general population is reported to be 67%, occurring more frequently in women than in men. Aging or other factors may be related to intrinsic degeneration associated with tendinopathy. The frequency of occurrence increases with age, leading to significant social participation and healthcare costs.

Shoulder pain and progressively increasing restriction of shoulder joint movement cause a reduction in shoulder joint positional awareness, upper extremity function, and quality of life. Losses in shoulder function affect individuals in many daily life skills, especially activities of daily living. The pain phenomenon that occurs during shoulder movements is the primary reason for these losses. Following this pain phenomenon, fear of movement or avoidance of movement may occur, leading to kinesiophobia.

In individuals with rotator cuff syndrome, there are not only functional impairments but also psychological impairments. The concept of "Psychological Resilience," which is among the psychological factors, is known to affect overall well-being. Especially in cases of persistent chronic shoulder pain, thoughts such as hopelessness and stress have a significant impact on psychosocial status. Psychosocial factors are thought to be quite effective in the severity of patients' pain and restrictions in joint range of motion. The literature indicates that individuals with high musculoskeletal pain have a high prevalence of anxiety and depression, particularly in chronic pain patients, and that psychological factors should be addressed.

The fear of movement and injury created by kinesiophobia is often followed by movement disorders and depression. It has been reported that individuals with high levels of kinesiophobia will avoid movement due to expecting the disease's course to worsen or for new symptoms to arise. Excessive avoidance of movement will lead to physical limitations in the individual's daily life. Consequently, a reduction in the patient's functionality will be observed. High psychological resilience has been found to be associated with lower pain severity, reduced joint limitations, and lower levels of kinesiophobia.

In physiotherapy, the dual definition of basic body awareness has been made. The first is the experience of the body (experiential dimension), and the second is movements and behaviors (movement dimension). In the context of physiotherapy, another definition of body awareness is the awareness of how the body is used in terms of its function, behavior, self, and interaction with others. Various sensory systems such as proprioception, interoception, exteroception, and the vestibular system are significant in the foundation of body awareness. For body awareness, the processing of interoceptive (sensory inputs coming from within the body) and exteroceptive (processing of inputs coming from outside the body) senses is necessary. Individuals' body awareness is related to movement capacity in daily life activities, health-related quality of life, body image, and pain severity findings.

While chronic basic body awareness has been studied in conditions like mental health, stroke, and chronic musculoskeletal problems, there are no studies examining basic body awareness in shoulder rehabilitation. Considering that psychological factors also affect the etiology of shoulder pain, our study aims to investigate the effect of basic body awareness level on shoulder functionality and psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of partial supraspinatus rupture by an orthopedics and traumatology specialist
* Shoulder pain lasting more than 4 weeks
* Unilateral shoulder pain,
* Not having been previously included in any physiotherapy program due to a shoulder problem,
* Body mass index (BMI) ≤ 30 kg/m²
* Individuals being cooperative

Exclusion Criteria:

* Having had shoulder surgery before,
* Receiving local corticosteroid injection/corticosteroid treatment within the last three months,
* Presence of uncontrolled neurological, cardiac, systemic disease that will prevent function,
* Presence of disease that will affect the cognitive and visual systems.

Inclusion Criteria for Healthy Volunteer Group

* Individuals between the ages of 30-65
* Healthy volunteer participants
* Participants of the same age and gender

Exclusion Criteria for Healthy Volunteer Group

* Presence of shoulder pain in the last 6 months
* Pain in 90° shoulder abduction and flexion
* Presence of night pain in the shoulder
* Having a body mass index (BMI) >30 kg/m2
* Having any systemic, neurological or rheumatological disease

Ages: 30 Days to 65 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 20 participants aged 30-65 years with rotator cuff tendinopathy who meet the inclusion criteria, along with 25 healthy volunteers of the same age and gender, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-02-22 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Baseline
  Pain Severity rated their feelings of pain on the line by themselves, thereby quantifying the pain.sual Analogue Scale Participants pain intensities ranged from "0" (no pain) to "10" (unbearable pain) to 10 cm will be evaluated with the Visual Pain Scale. The pain intensity of the participants before and after the treatment was evaluated at rest and during activity.
Evaluation of joint range of motion | Baseline
  Baseline digital Absolute + Axis goniometer device will be used. Flexion, extension, abduction, internal and external rotation range of motion of the shoulder joint will be evaluated in degrees. For each joint range of motion value, 3 consecutive measurements will be taken and the average value will be recorded.
American Shoulder and Elbow Surgeons (ASES) | Baseline
  American Shoulder and Elbow Surgeons (ASES) created the ASES questionnaire in order to develop a standardized method for evaluating shoulder function. The goal was to design a questionnaire that was easy to use, assessed function, and was entirely based on patient self-evaluation. The ASES score totals 100 points and allocates 50 points for measuring function and 50 points for pain.
Body Awareness Questionnaire | Baseline
  The body awareness questionnaire is a 18 item scale, with the total scale score calculated as a sum of the items.
  Items are scored on a 1-7 scale, with the total scale score calculated as a sum of the items. The questions with asterisks are reverse scored. This means that for example, if someone scored 1 it would now be a score of 5.
Body Image Survey (BIA) | Baseline
  BIA was used to measure the patients' level of satisfaction with their body image. BIA consists of a person's body parts or functions.It is a scale that determines satisfaction. It was shown in the study by Hovardaoğlu et al. that the scale is valid and reliable in Turkish.
Rotator Cuff Quality of Life | Baseline
  It is a questionnaire that evaluates the quality of life in rotator cuff injuries. It is a disease-specific questionnaire and is distinctive in assessing quality of life. It is a questionnaire consisting of 34 questions and 5 subparameters that evaluates the physical symptoms of the disease, work activities, daily living activities, social and emotional status. Each question is calculated out of 100 points and the total score is expressed as a percentage.
The Tampa Scale for Kinesiophobia (TSK) | Baseline
  The Tampa Scale for Kinesiophobia (TSK) is a self-report questionnaire that is used to assess an individual's fear of movement or re-injury. The TSK consists of 17 items that ask respondents to rate their level of agreement with statements related to the fear of movement or re-injury. A high score from the scale indicates a high level of kinesiophobia.
Assessment of Anxiety and Depression | Baseline
  The participants' anxiety and depression levels will be assessed with the Hospital Anxiety and Depression Scale.The scale was developed by Zigmond and Snaith to assess anxiety and depression levels. 7 of the 14 questions assess anxiety and 7 assess depression. Each item is scored between 0 and 3. High scores obtained from the scale indicate high anxiety and depression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, PhD, Study Director — Medipol University
Locations (1):
- Özlem Görgülü Göksu, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No